CLINICAL TRIAL: NCT07379944
Title: The Effect of Guided Visualization Meditation on Surgical Stress Response in Patients Undergoing Cardiac Surgery: A Nonrandomized Controlled Clinical Trial
Brief Title: Guided Visualization Meditation for Reducing Surgical Stress Response in Cardiac Surgery Patients
Acronym: GVM-CARDIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Tuğba Albayram, Research Assistant Dr, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/358
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery; Surgical Stress Response; Coronary Artery Disease; Postoperative Stress; Anxiety
Keywords: guided visualization; meditation; mind-body intervention; STAI; perioperative care; cardiac surgery patients; insulin resistance; blood glucose
MeSH Terms: conditions — Coronary Artery Disease; Anxiety Disorders; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Nonrandomized, parallel-group clinical trial evaluating the effects of guided visualization meditation compared with standard care in patients undergoing cardiac surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Visualization Meditation (Experimental): A 15-20 minute guided visualization audio session including verbal imagery and relaxation techniques. Delivered via headphones twice daily on the preoperative day, surgery day, and postoperative day 1.
  Interventions: Behavioral: Guided Visualization Meditation
- Standard Care (No Intervention): Participants receive routine perioperative standard care without guided visualization meditation. All biometric and psychological measurements are collected at the same time points as the intervention group.

INTERVENTIONS:
Behavioral: Guided Visualization Meditation — A 15-20 minute guided visualization audio session including verbal imagery and relaxation techniques. Delivered via headphones twice daily on the preoperative day, surgery day, and postoperative day 1.
  Arms: Guided Visualization Meditation

SUMMARY:
This study aims to evaluate whether guided visualization meditation can reduce the surgical stress response in patients undergoing open-heart surgery. Surgical stress response includes changes in hormones, blood glucose, and anxiety levels that occur before and after major surgery. Guided visualization meditation is a non-invasive relaxation technique that uses calming audio instructions to help patients imagine peaceful scenes and reduce stress.

In this study, patients scheduled for cardiac surgery will be assigned to one of two groups: an intervention group that receives guided visualization meditation and a control group that receives standard care only. Patients in the intervention group will listen to an audio recording containing guided visualization and calming background music through headphones. Sessions will be provided twice on the day before surgery, twice on the day of surgery, and twice on the first postoperative day.

To evaluate the effects of the intervention, blood samples will be collected to measure cortisol, glucose, and insulin levels. Anxiety levels will be assessed using the State-Trait Anxiety Inventory (STAI-I and STAI-II), and pain will be measured using a visual pain scale. These measurements will be performed at three specific time points: one day before surgery, six hours after extubation, and one day post-surgery.

The goal of this research is to determine whether guided visualization meditation can help reduce stress-related physiological and psychological changes in patients undergoing cardiac surgery. If effective, this method may offer a simple, safe, and supportive strategy to improve recovery and overall patient well-being.

DETAILED DESCRIPTION:
Major cardiac surgery triggers a strong neuroendocrine and psychological stress response, which can negatively affect postoperative recovery. The surgical stress response is primarily characterized by increased cortisol secretion, elevated blood glucose levels, insulin resistance, fluid retention, increased cardiac workload, and heightened anxiety. Excessive or prolonged stress response may contribute to complications, delayed healing, and extended intensive care or hospital stay. Reducing the magnitude of the surgical stress response is considered an important component of perioperative patient management.

Guided visualization meditation is a non-pharmacologic mind-body technique that uses structured verbal guidance, calming metaphors, and controlled breathing cues to help individuals focus attention on peaceful imagery. This technique may influence autonomic nervous system activity, reduce sympathetic arousal, and improve emotional regulation. Prior studies suggest that guided relaxation strategies can lead to reductions in cortisol, improvements in anxiety levels, and improved patient comfort. However, there is limited evidence regarding their effectiveness in patients undergoing open-heart surgery.

This study is designed as a non-randomized, controlled, interventional clinical trial with two parallel groups: an intervention group receiving guided visualization meditation and a control group receiving standard postoperative care. Each participant in the intervention group will listen to a 15-20 minute guided visualization audio recording with calming background music twice daily on three consecutive days: the day before surgery (T0), the day of surgery (T1), and the first postoperative day (T2). Audio will be delivered through headphones in a quiet clinical environment.

Primary outcomes will include serum cortisol levels measured at T0, T1 (six hours after extubation), and T2. Secondary outcomes will include serum glucose and insulin levels, State-Trait Anxiety Inventory scores (STAI-I and STAI-II), and pain scores assessed using a visual pain scale. All biochemical samples will be obtained by clinical staff following routine safety protocols. Anxiety and pain assessments will be completed face-to-face by trained research personnel.

Eligibility criteria include adults aged 18 or older scheduled for first-time on-pump cardiac surgery via median sternotomy, ASA I-II classification, mild to moderate hypothermia protocol, and the absence of psychiatric diagnoses or corticosteroid use. Patients experiencing complications, prolonged surgery, or altered postoperative consciousness will be excluded.

Data will be collected prospectively and analyzed using statistical software (SPSS). Descriptive statistics, normality testing, and appropriate comparative tests (ANOVA, repeated-measures analyses) will be applied to evaluate changes over time and differences between groups. The primary hypothesis is that guided visualization meditation will result in significantly lower cortisol levels and reduced anxiety compared to standard care.

This research aims to contribute to supportive care practices in cardiac surgery by evaluating a low-cost, non-invasive, and easily implementable intervention that may help regulate neuroendocrine stress responses and improve postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled to undergo open-heart surgery
* ASA physical status I-II
* First-time cardiac surgery
* On-pump, median sternotomy technique planned
* Mild to moderate intraoperative hypothermia protocol
* No diagnosed psychiatric disorder
* Not using psychotropic medications
* No endocrine disorders affecting cortisol (e.g., Addison's disease, Cushing's syndrome)
* Not taking corticosteroid medications
* Glasgow Coma Score = 15 postoperatively
* No perioperative complications that may interfere with participation
* Able and willing to provide informed consent

Exclusion Criteria:

* Prolonged or complicated surgery
* Withdrawal of consent at any stage
* Postoperative altered consciousness (GCS < 15)
* Perioperative administration of corticosteroids
* Severe intraoperative complications
* Surgery cancelled or rescheduled
* Hearing impairment preventing participation in auditory intervention
* Any condition clinically judged by the investigator to interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Serum Cortisol Level | One day before surgery, six hours after extubation on the day of surgery, and one day after surgery
  Serum cortisol levels will be measured at three perioperative time points to evaluate the neuroendocrine surgical stress response. A reduction in cortisol levels in the intervention group compared with the control group will indicate the effectiveness of guided visualization meditation.

SECONDARY OUTCOMES:
Serum Glucose Level | One day before surgery, six hours after extubation on the day of surgery, and one day after surgery
  Serum glucose levels will be measured at three perioperative time points to assess
Serum Insulin Level | One day before surgery, six hours after extubation on the day of surgery, and one day after surgery
  Serum insulin levels will be measured to evaluate perioperative insulin resistance as part of the surgical stress response. Lower insulin levels in the intervention group compared with the control group will suggest improved metabolic stability.
State Anxiety (STAI-S) State Anxiety Score Measured by the State-Trait Anxiety Inventory (STAI-S) | One day before surgery, six hours after extubation on the day of surgery, and one day after surgery
  State anxiety will be assessed using the State-Trait Anxiety Inventory - State Form (STAI-S). The scale ranges from 20 to 80, with higher scores indicating higher anxiety levels. Lower scores in the intervention group will reflect reduced situational anxiety.
Trait Anxiety (STAI-T) | One day before surgery and one day after surgery
  Trait anxiety will be assessed using the State-Trait Anxiety Inventory - Trait Form (STAI-T). The scale ranges from 20 to 80, with higher scores indicating higher anxiety levels. A reduction in scores after surgery will indicate decreased persistent anxiety.
Pain Score (VAS) | One day before surgery, six hours after extubation on the day of surgery, and one day after surgery
  Pain will be evaluated using the Visual Analog Pain Scale, ranging from 0 to 10, where higher scores indicate more severe pain. Differences between groups will determine whether guided visualization meditation contributes to postoperative pain relief.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to patient privacy protections, ethical committee restrictions, and institutional data confidentiality policies. Only aggregated statistical results will be made available upon reasonable request.